CLINICAL TRIAL: NCT05180721
Title: A Multi-level Intervention to Increase Access and Use of the Patient Portal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000031753; R21MD016949-01 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-01-06 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Patient Education; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of patient portal for diabetes management (Experimental): A multi-level intervention aimed at increasing access and use of patient portals for diabetes management (MAP) in community health centers (CHCs).
  Interventions: Behavioral: Use of patient portal for diabetes management

INTERVENTIONS:
Behavioral: Use of patient portal for diabetes management — A multi-level intervention aimed at increasing access and use of patient portals for diabetes management (MAP) in community health centers (CHCs).

SUMMARY:
The purpose of the study is to develop and evaluate a multi-level intervention aimed at increasing access and use of patient portals for diabetes management (MAP) in community health centers (CHCs).

DETAILED DESCRIPTION:
Prior to the clinical trial, qualitative methods were used to inform the intervention protocol. For the clinical trial, a pilot study will be conducted to evaluate the effect of the intervention on patient portal use, patient engagement with care, and clinical outcomes in adults with type 2 diabetes. The focus of this registration is the clinical trial.

Using a within subjects, pre-post design the investigator will pilot MAP in an anticipated 30 adults with T2D who are not using the portal. Data will be collected at baseline, 3, and 6 months. The investigators will evaluate the feasibility of MAP using an established framework (acceptability, demand, implementation, adaptation, and integration.

The intervention will consist of the following:

1. provide free access to tablets and internet (material circumstances);
2. technology training and ongoing support (psychosocial factors);
3. assess social determinants of health and refer to community resources (material circumstances);
4. support diabetes self-management behaviors and refer to clinic services (behavioral and biological factors).

MAP will be delivered by community health workers (CHW) and nurses already embedded in CHCs (healthcare system). The 3-month intervention is thoughtfully sequenced to first have CHWs address patient portal access (tablet, home internet), and then move on to patient mastery of the tablet and portal functionality. Next, CHWs will assess social determinants of health using an established measure and connect the participant to relevant community resources (e.g., SNAP benefits). It is anticipated that participants will have 4-6 individual sessions with the CHW, approximately 30 minutes each, followed by ongoing technology support as needed.

Next, the clinic nurse will proactively contact the participant via the portal to provide diabetes self-management support. The nurse will begin by assessing participant behaviors and will then work with the participant to co-create a plan to help with diabetes self-management. The plan will include referral to relevant ancillary clinic services as needed (e.g., DSM education [DSME], nutritionist, obtaining a glucose meter). Participants will be instructed and encouraged to upload blood glucose data and communicate with the nurse and their health care provider via the portal, both of which have been shown to improve glycemic control. The nurse will work with each patient to individualize DSMS behavioral targets, considering the following priorities: use of the portal, attendance at appointments, uploading of blood glucose data to the portal, medication refills and adherence, and lifestyle and emotional factors. It is anticipated that nurses will communicate with patients via the portal at least twice weekly during the first month followed by ongoing DSMS as needed. In-person or telehealth sessions will be scheduled as needed. However, the exact sequence, timing, and length of sessions will be participant driven. For example, a participant who learns the portal quickly may proceed at a faster rate, or a participant who already uploads glucose data may skip that step.

ELIGIBILITY:
Inclusion Criteria:

* Established patient of one of the partner CHCs
* Age > 18 years
* Diagnosed with T2D >6 months
* Able to read in English or Spanish
* Not using the patient portal
* A1c >7.5%

Exclusion Criteria:

* Cognitive impairment (≥3 errors on the Six Item Screener for cognitive impairment in clinical research [SIS]) (Callahan et al. 2002) as they will have difficulty in completing the study requirements
* Gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whittemore, PhD, APRN, Study Chair — Yale University
Locations (2):
- United States (2):
  - Fair Haven Community Health Center, New Haven, Connecticut
  - Norwalk Community Health Center, Norwalk, Connecticut

REFERENCES:
- [Derived] Wagner J, Akyirem S, Lipson J, Chen HN, Whittemore R. Evaluation of the implementation of a patient portal pilot intervention among people with type 2 diabetes at community health centers. Front Clin Diabetes Healthc. 2026 Jan 6;6:1689830. doi: 10.3389/fcdhc.2025.1689830. eCollection 2025. PMID 41567495
- [Derived] Whittemore R, Jeon S, Akyirem S, Chen HNC, Lipson J, Minchala M, Wagner J. Multilevel Intervention to Increase Patient Portal Use in Adults With Type 2 Diabetes Who Access Health Care at Community Health Centers: Single Arm, Pre-Post Pilot Study. JMIR Form Res. 2025 Mar 25;9:e67293. doi: 10.2196/67293. PMID 40131327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two community health centers. Flyers were posted in the clinics. Clinic personnel identified potentially eligible participants and if interested, would refer to research team. A trained research assistant provided information about the study and obtained informed consent in the preferred language of participant (Spanish or English).
Groups:
- Use of Patient Portal for Diabetes Management: A multi-level intervention aimed at increasing access and use of patient portals for diabetes management (MAP) in community health centers (CHCs).
  1. Provision of table and 6 month data plan for internet
  2. Technology training
  3. Diabetes support
  4. Text message/phone calls
Period: Overall Study
Arm/Group | Use of Patient Portal for Diabetes Management
Started | 26
Completed | 22
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: There were 4 participants lost to follow-up so their data was not included in our final report. They were not exposed to any aspect of the intervention.
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.32 (10.93)

OUTCOME MEASURES:

1. Primary Outcome: Usage of Portal
Description: Frequency. Mean portal login days/per month will be calculated using the EMR system
Time Frame: Monthly for 6 months
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
days per month
  Mean of first 3 months | 12.65 (6.21)
  Mean of 3- 6 months | 5.79 (3.74)

2. Primary Outcome: Change in A1C Value
Description: The A1C value will be assessed via fingerprick point of care A1c kits.
Time Frame: Baseline, 3 months and 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
percent
  Baseline | 8.31 (1.65)
  3 months | 8.09 (1.64)
  6 months | 8.23 (1.35)

3. Secondary Outcome: Summary of Self-Care in Diabetes Survey- Diet
Description: Diet - following diabetes diet over past 7 days (score range 0-7, with higher scores indicating better self-care)
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
score on a scale
  Baseline | 2.82 (2.91)
  3 months | 4.00 (2.54)
  6 months | 3.68 (2.80)

4. Secondary Outcome: Diabetes Self-Efficacy
Description: Self-confidence in diabetes self-management tasks (score range from 1-5 with higher scores indicating better diabetes self-efficacy)
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
score on a scale
  Baseline | 3.14 (1.01)
  3 months | 3.44 (1.17)
  6 months | 3.68 (2.80)

5. Secondary Outcome: Health Care Climate Questionnaire
Description: Perception of support by health care providers with higher scores indicating more perceived support, scores range from 1-5
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
score on a scale
  Baseline | 4.15 (0.78)
  3 months | 4.14 (0.83)
  6 months | 3.95 (1.07)

6. Secondary Outcome: Problem Areas in Diabetes (PAID)
Description: Score ranges from 0-100 with higher scores indicating more distress
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of Patient Portal for Diabetes Management
Number analyzed (Participants) | 22
score on a scale
  Baseline | 43.58 (30.51)
  3 months | 29.09 (23.03)
  6 months | 25.45 (24.88)

ADVERSE EVENTS:
Time Frame: From enrollment to approximately 6 months
Arm/Group | Use of Patient Portal for Diabetes Management
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT05180721/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05180721/ICF_001.pdf